CLINICAL TRIAL: NCT02186119
Title: A Study of Abicipar Pegol in Patients With Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 150998-004; PALM (Other: Allergan)
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — abicipar pegol; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- abicipar pegol 2 mg (group A) (Experimental): Abicipar pegol 2 mg administered to the study eye by intravitreal injection at day 1, weeks 4, 8, and 20, followed by a sham procedure at weeks 12, 16, and 24.
  Interventions: Drug: abicipar pegol; Other: sham procedure
- abicipar pegol 2 mg (group B) (Experimental): Abicipar pegol 2 mg administered to the study eye by intravitreal injection at day 1, weeks 4, 8, 16, and 24, followed by a sham procedure at weeks 12 and 20.
  Interventions: Drug: abicipar pegol; Other: sham procedure
- abicipar pegol 1 mg (Experimental): Abicipar pegol 1 mg administered to the study eye by intravitreal injection at day 1, weeks 4, 8, 16, and 24, followed by a sham procedure at weeks 12 and 20.
  Interventions: Drug: abicipar pegol; Other: sham procedure
- ranibizumab (Active Comparator): Ranibizumab (Lucentis®) administered to the study eye by intravitreal injection every 4 weeks from day 1 through week 24.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: abicipar pegol — Abicipar pegol administered to the study eye by intravitreal injection at the visits noted per protocol.
  Arms: abicipar pegol 1 mg; abicipar pegol 2 mg (group A); abicipar pegol 2 mg (group B)
Drug: ranibizumab — Ranibizumab (Lucentis®) administered to the study eye by intravitreal injection every 4 weeks from day 1 through week 24.
  Other Names: Lucentis®
  Arms: ranibizumab
Other: sham procedure — Sham procedure to the study eye at the visits noted per protocol.
  Arms: abicipar pegol 1 mg; abicipar pegol 2 mg (group A); abicipar pegol 2 mg (group B)

SUMMARY:
This is a safety and efficacy study of abicipar pegol in patients with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus (Type 1 or 2)
* Decreased vision due to diabetic macular edema in at least 1 eye
* Best corrected visual acuity of 20/32 to 20/320 in the study eye and 20/200 or better in the fellow eye

Exclusion Criteria:

* Stroke or heart attack within the past 3 months
* History of vitrectomy, macular surgery, or glaucoma surgery in the study eye
* Cataract or refractive surgery in the study eye within the last 3 months
* Laser photocoagulation of the study eye within the last 3 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Best Corrected Visual Acuity (BCVA) | Baseline, Week 28

SECONDARY OUTCOMES:
Percentage of Patients with a BCVA Gain of ≥15 Letters in the Study Eye on the Early Treatment Diabetic Retinopathy Study (ETDRS) Scale | Baseline, 28 Weeks
Change from Baseline in Central Retinal Thickness (CRT) in the Study Eye | Baseline, Week 28
Percentage of Patients with a BCVA of ≥70 Letters | 28 Weeks
Percentage of Patients with Resolution of Macular Edema | 28 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- United States (2):
  - Gilbert, Arizona
  - Abilene, Texas